CLINICAL TRIAL: NCT03501095
Title: Evaluation of Laryngeal Morbidity After Orotracheal Intubation by Vocal Analysis and Laryngostroboscopy: A Pilot Study
Brief Title: Evaluation of Laryngeal Morbidity After Orotracheal Intubation by Vocal Analysis and Laryngostroboscopy
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Rosanna Vaschetto, MD, PhD, medical physician, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: AOCarita
Record Dates: First submitted 2018-03-07; First posted 2018-04-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Intubation Complication; Vocal Cord Dysfunction; Vocal Tone Disorder; Intubation;Difficult
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: patients who must undergo general and/or urology surgery of an elective type
  Interventions: Diagnostic Test: Vocal analysis and Laryngostroboscopy

INTERVENTIONS:
Diagnostic Test: Vocal analysis and Laryngostroboscopy — Vocal analysis study the acoustic emission of the pneumo-phono-articulatory system, i.e. the vocal signal. Currently, digital technology instruments enable the processing and analysis of the verbal signal quickly and reliably, also offering graphical products and numerical data. Among the various existing software products for the study of the vocal signal, PRAAT is available. In practice, the vocal parameters are acquired in a non-invasive way with a microphone.
  Laryngostroboscopy is one of the most widely used techniques for laryngeal clinical evaluation. This is a non-invasive endoscopic practice performed by means of a flexible fibroscope, which, through a pulsed light source, allows visualization of the chordal movement.
  Other Names: Vocal analysis; Laryngostroboscopy

SUMMARY:
The delicate structures of the larynx can be compromised by innumerable causes, one of these is represented by endotracheal intubation. More frequently, these damages are represented by hematomas, edema and granulomas of the vocal cords. The pathophysiology of laryngeal damage can be explained by an ischemic attack of the chordal mucosa. Numerous risk factors can cause the onset of damage, some depending on the practice itself, such as size and type of endotracheal tube, cuff pressure, use of mandrels and / or inserting devices, use of oral or nasogastric tubes, use of neuromuscular inhibitors or sleep-inducing drugs and the duration of the intervention; others from patient-related factors, such as gender, weight, history of exposure of smoking habit, or a history of gastroesophageal reflux (GERD). The incidence of such symptoms varies from 0% to 18% among the general population, with an average of 6% with resolution of most of the symptoms within 72 hours unless substantial damage has occurred to the vocal cords or to the arytenoids. In general, the incidence of such laryngeal complications has been described by several studies, but there is no standardized protocol for measuring and evaluating their entity. The purpose of this study is to determine how the voice and the chordal clinical aspect vary after oro-tracheal intubation, evaluated through voice analysis and laryngostroboscopy.

DETAILED DESCRIPTION:
Acoustic analysis aims at studying the acoustic emission of the pneumo-phono-articulatory system, i.e. the vocal signal. Currently, digital technology instruments enable the processing and analysis of the verbal signal quickly and reliably, also offering graphical products and numerical data. Among the various existing software products for the study of the vocal signal, PRAAT is available.

In practice, the vocal parameters are acquired in a non-invasive way with a microphone. At the same time, these analysis systems can be integrated by other methods, such as laryngostroboscopy. This method is one of the most widely used techniques for laryngeal clinical evaluation. This is a non-invasive endoscopic practice performed by means of a flexible fibroscope, which, through a pulsed light source, allows visualization of the chordal movement.

At first, a study will be carried out on healthy volunteers, comparable for their demographic characteristics to the second population to be included. In this way the investigators will test the instrument used for the voice analysis, in order to set the reference values for the general population. In a second step, the investigators will evaluate the incidence of post-intubation laryngeal complications, considering as a pathological all values above 95% percentile compared to healthy individuals.

During the first phase, healthy volunteers will undergo voice analysis in two different days. Subsequently, the patients included in the study population will be undergo during the preoperative, intraoperative and postoperative to a combined evaluation between Anesthesiologists and ENTs for data collection.

The data to be recorded, both for the healthy volunteers as well as for patients, will include personal data, anamnestic, working exposure and specific risk factors such as smoking, alcohol, irritants, a previous diagnosis of GERD, frequent inflammation of upper respiratory tract (VADS); moreover, only for patients, the pre-, intra and post-surgery anesthesia evaluation parameters will be collected.

During the pre-surgery visit, patients will receive an otorhinolaryngeal evaluation by laryngostroboscopy and the vocal analysis.

Any lesions due to endotracheal intubation will be standardized according to Mendels et al.'s modified classification, in grade I (lesion of the vocal cords in terms of vibratory changes, which can be observed in the epithelium, lamina propria or arytenoid cartilages ) and grade II (vocal cords movement disorders in terms of paralysis, arytenoid dislocation or incomplete glottal closure).

The vocal analysis will consist, instead, in asking the patient to voice through a microphone (Sennheiser E 835 S) placed at about 15 cm from the mouth, a certain vowel (ie "a") and recording it using PRAAT software (version 6.0. 29 64bit). The PRAAT is a multi-platform application developed since 1992, constantly updated and made available free of charge by Paul Boersma and David Wenink of the Phonetics Laboratory of the University of Amsterdam. It provides numerical data with the possibility of objective evaluations of the vocal characteristics. The system provides information on the fundamental frequency (F0), glottal impulses, microperturbations or causal variations of the fundamental period (Jitter) and of the amplitude (Shimmer) and also the relationship between the periodic and aperiodic signal (NHR).

F0 is the frequency of vocal cord vibrations during phonation, it is calculated in Hz and it differs from man to woman with a difference of about 1.5 times higher in women.

Jitter is a parameter related to the microperturbation of the fundamental period and in particular the Jitter % represents the percentage ratio between the absolute average of the differences between the consecutive fundamental periods and the average fundamental period. The parameters relating to changes in the fundamental period increase in the presence of an irregular glottal vibration.

The Shimmer identifies the microperturbations of the signal amplitude, therefore the Shimmer % expresses the average relative perturbation of the amplitude period; the values increase in case of organic or functional vocal pathology, as a consequence of the inability of the chordal oscillator to maintain a regular vibration.

NHR (noise-to-harmonics ratio) expresses the relationship between the disharmonic component (noise) and the harmonic component, it constitutes a global evaluation of the presence of noise in the analyzed signal due to the simultaneous variation of frequency and amplitude, of turbulent noise, of sub-harmonic components and sound interruptions; its increase is related to the subjective perception of dysphonia.

Then, after a forced inhalation, the sound emitted until exhaustion will represent the maximum phonatory time (MPT), ie the longest time during which a patient can sustain the phonation of a vowel sound and it is calculated in seconds (s). These measurements will be performed three consecutive times; for the F0 variation, Jitter %, Shimmer % and NHR will be kept the avarage value while for the MPT the best recording will be kept.

Finally, the investigators will submit to the subject a self-assessment questionnaire on the quality of the voice (Voice Handicap Index or VHI 10). This assessment is necessary to estimate the psychological and social impact of the severity of dysphonia according to the subject with regard to his normal daily activity. In this case, it will help the investigators to exclude patients with pre-existing dysphonic problems. It will not be used after surgery, since it is not indicative of short term variations. The anaesthesiological evaluation will consist of a normal pre-surgery visit with particular regard to demographic and anamnestic parameters and difficulties associated with respiratory tract, which will be indicated in the appropriate form.

During surgery patients will be monitored and the respiratory tract will be handled as the usual standard of care, collecting all necessary data for subsequent evaluations. 24-48 hours after surgery, the patient, still hospitalized, will undergo an otorhinolaryngeal re-evaluation by means of vocal analysis and laryngostroboscopy.

In case of laryngeal morbidity (i.e edema, granulomas, mucosal damage, cordial paralysis and/or alterations in the voice characteristics) the patient will be advised to undergo an otorhinolaryngology visit.

The pilot study will enroll patients who must undergo general and/or urology surgery of an elective type.

ELIGIBILITY:
Inclusion Criteria:

* all patients between the age of 18 and 70 years old who have given informed consent and who must undergo general or urological surgery will be included.

Exclusion Criteria:

* age: below 18 or over 70 years old,
* refusal of the patient to consent,
* risk of the American Society Anesthesiologists (ASA) > III,
* patients previously subjected to demolition surgery of head-neck and/or chemo-radiotherapy of the same structures,
* patients with a history of hoarseness, vocal tract abnormalities and / or hearing impairment.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators will study patients undergoing general anesthesia for urological or general surgery at the University Hospital (AOU) Maggiore della Carità di Novara in the time span between 1st April 2018 to 31st March 2019.
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence, expressed as the number of new cases per year, of laryngeal complications arising after endotracheal intubation. This complications will be related to: | Presence of laryngeal damage 24-48 hours after surgery not visible at the pre-surgery visit.
  1. the variation of voice parameters, during acoustic analysis, above 95% percentile, compared to healthy volunteers, of patients who undergo orotracheal intubation.
  2. the presence or absence of laryngeal damage at laryngostroboscopy.

SECONDARY OUTCOMES:
Correlation between weight and modified Mallampati | The data will be assessed during pre-surgery visit
  On the x axis will be plotted the weight measured in kilograms, on y axis will be plotted Mallampati scale.
Correlation between endotracheal tube size and presence of laryngeal damage | The data will be assessed 24 hours after surgery
  the size tube is measured in millimeters while laryngeal damage will be measured by Mendel's scale
Correlation between use or not of mandrel and the modifications of Jitter % | The data will be assessed 24 hours after surgery
  The Jitter % will be measured with software PRAAT
Correlation between use or not of mandrel and the modifications of Shimmer % | The data will be assessed 24 hours after surgery
  The Shimmer % will be measured with software PRAAT

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mota LA, de Cavalho GB, Brito VA. Laryngeal complications by orotracheal intubation: Literature review. Int Arch Otorhinolaryngol. 2012 Apr;16(2):236-45. doi: 10.7162/S1809-97772012000200014. PMID 25991942
- [Background] Mendels EJ, Brunings JW, Hamaekers AE, Stokroos RJ, Kremer B, Baijens LW. Adverse laryngeal effects following short-term general anesthesia: a systematic review. Arch Otolaryngol Head Neck Surg. 2012 Mar;138(3):257-64. doi: 10.1001/archoto.2011.1427. PMID 22431870
- [Background] Maktabi MA, Smith RB, Todd MM. Is routine endotracheal intubation as safe as we think or wish? Anesthesiology. 2003 Aug;99(2):247-8. doi: 10.1097/00000542-200308000-00002. No abstract available. PMID 12883393
- [Background] Horii Y, Fuller BF. Selected acoustic characteristics of voices before intubation and after extubation. J Speech Hear Res. 1990 Sep;33(3):505-10. doi: 10.1044/jshr.3303.505. PMID 2232768
- [Background] Peppard SB, Dickens JH. Laryngeal injury following short-term intubation. Ann Otol Rhinol Laryngol. 1983 Jul-Aug;92(4 Pt 1):327-30. doi: 10.1177/000348948309200402. PMID 6881831
- [Background] Beckford NS, Mayo R, Wilkinson A 3rd, Tierney M. Effects of short-term endotracheal intubation on vocal function. Laryngoscope. 1990 Apr;100(4):331-6. doi: 10.1288/00005537-199004000-00001. PMID 2319880
- [Background] Hamdan AL, Sibai A, Rameh C, Kanazeh G. Short-term effects of endotracheal intubation on voice. J Voice. 2007 Nov;21(6):762-8. doi: 10.1016/j.jvoice.2006.06.003. Epub 2006 Aug 14. PMID 16905292